CLINICAL TRIAL: NCT05149768
Title: An Open Label Extension Study of Brentuximab Vedotin Treatment in Active Diffuse Cutaneous Systemic Sclerosis (Diffuse Scleroderma)
Brief Title: Open Label Extension Study of Brentuximab Vedotin in Early dcSSc
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Seattle Genetics (now a wholly owned subsidiary of Pfizer) (Unknown); Pfizer (Industry)
Responsible Party: Principal Investigator, Janet Pope, Head of Rheumatology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BV202108
Record Dates: First submitted 2021-11-24; First posted 2021-12-08 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; brentuximab vedotin; CD30-directed antibody-drug conjugate; antirheumatic agents; antineoplastic agents; skin diseases; immunologic factors
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Skin Diseases | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Administration of Brentuximab vedotin (Experimental): Maximum duration of treatment: 48 weeks Maximum dose allowed: 0.6 mg/kg Route of administration: intravenous
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — Dose 0.6mg/kg will be given every 3 weeks for 16 cycles (48 weeks), in addition to standard of care medications for SSc that may include cyclophosphamide, methotrexate, azathioprine, mycophenolate mofetil (MMF, cellcept) and mycophenolic acid (myfortic)
  Other Names: ADCETRIS, SGN-35

SUMMARY:
The purpose of this study is to assess safety and efficacy of Brentuximab vedotin, a CD30-directed antibody-drug conjugate, in patients with active diffuse cutaneous systemic sclerosis (dcSSc) who relapsed after discontinuation of Brentuximab vedotin.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc, Scleroderma) is a multisystem autoimmune disease characterized by widespread vascular injury and progressive fibrosis of the skin and internal organs. Internal organ involvement results in increased mortality of SSc patients. There is no effective treatment for the majority of patients with early active diffuse scleroderma (diffuse cutaneous systemic sclerosis; dcSSc). It's possible to reverse immune inflammation and reduce the probability of irreversible fibrosis early in the disease course via significant immune modulation. The preliminary results of the Phase II study of Brentuximab vedotin (Protocol BV201708) in SSc demonstrated the short-term safety and benefits of this treatment as many participants already achieved the primary endpoint at 24 weeks. This study is proposed as an extension of the ongoing protocol for up to 48 weeks to make the treatment available for SSc patients who have significantly improved on Brentuximab vedotin, but relapsed after discontinuation of the treatment. Similar to the ongoing Phase II study, the Health Assessment Questionnaire Disability Index (HAQ-DI), patient and physician global scores, inflammatory markers (ESR, CRP), and combined response index in SSc (CRISS) and changes in CD30-stained cells on skin biopsies with IHC will all be exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diffuse cutaneous systemic sclerosis enrolled in the Phase II Adcetris study (BV201708) at St. Joseph's Health centre, aged 18 years or older, and:
2. Worsening mRSS of ≥ 4 points as compared to mRSS score at the end of treatment visit (week 48) in the initial study (BV201708).
3. Able to give informed consent.

Exclusion Criteria:

1. Poor pulmonary function (FVC<40% and/or DLCO<30%).
2. Pregnancy, breast feeding or child bearing potential without practicing highly effective contraception (and partners for men in the study).
3. Clinically significant pulmonary hypertension requiring drug therapy.
4. Clinically significant cardiac disease.
5. Chronic or ongoing active infectious disease requiring systemic treatment.
6. Seropositivity for human immunodeficiency virus (HIV).
7. Active tuberculosis (TB) infection.
8. Active viral infection with viral replication of hepatitis B or C virus.
9. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, pancreatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease; and cancer.
10. Peripheral neuropathy at screening Grade 2 or higher.
11. Known or suspected hypersensitivity to components of the treatment
12. Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
13. Any of the following laboratory abnormalities at screening:

    * Absolute neutrophils count <2.0 x 109/L
    * Hemoglobin <85 g/L
    * Platelet count < 100 x 109/L
    * AST/SGOT or ALT/SGPT >2.0 UNL
14. Participation in another clinical trial within six weeks before randomization in this study, with the exception of continuation from the initial study BV201708.
15. Use of rituximab within the previous 4 months.
16. Immunization with a live/ attenuated vaccine less than 4 weeks prior to the baseline visit.
17. Current or history of progressive multifocal leukoencephalopathy (PML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-02-14 (Actual); Primary Completion 2026-02-14 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in skin thickness measured by modified Rodnan Skin Score | 48 weeks
  Skin improvement is defined as the mean mRSS decrease of ≥8 points
  modified Rodnan Skin Score (mRSS): is a standard outcome measure for skin disease in SSc and calculated by measuring skin thickness in 17 different body sites (each site scored 0-3, with a total possible additive score of 51). A higher skin score (or a higher "skin thickness") and progression of this score, is predictive of internal organ involvement and mortality. While a lower or improving (lessening) score is associated with favorable outcomes, including better survival.

SECONDARY OUTCOMES:
Change in skin thickness over time measured by modified Rodnan Skin Score | 12 weeks and 36 weeks
  modified Rodnan Skin Score (mRSS): is a standard outcome measure for skin disease in SSc and calculated by measuring skin thickness in 17 different body sites (each site scored 0-3, with a total possible additive score of 51). A higher skin score (or a higher "skin thickness") and progression of this score, is predictive of internal organ involvement and mortality. While a lower or improving (lessening) score is associated with favorable outcomes, including better survival.
Change in physician global assessment of disease activity | 12, 24, 36, and 48 weeks.
  Measured on a Visual Analogue Scale (VAS) from 0-10, with 0 being no disease activity and 10 being the worst possible disease activity.
Change in physician global assessment of disease severity | 12, 24, 36, and 48 weeks
  Measured on a Visual Analogue Scale (VAS) from 0-10, with 0 being no disease severity and 10 being the worst possible disease severity.
Change in physician global assessment of disease damage | 12, 24, 36, and 48 weeks
  Measured on a Visual Analogue Scale (VAS) from 0-10, with 0 being no disease damage and 10 being the worst possible disease damage.
Change in patient global assessment of health status | 12, 24, 36, and 48 weeks
  Measured on a Visual Analogue Scale (VAS) from 0-100, with 0 being no overall effect of disease on participant, and 100 being the worst possible overall effect of disease on participant.
  This is a patient reported outcome.
Change in Scleroderma Health Assessment Questionnaire (SHAQ) | 12, 24, 36, and 48 weeks
  The SHAQ combines the disability and pain scales of the HAQ (HAQ-DI), with five scleroderma-specific Visual Analogue Scales for: digital ulcers, Raynaud's phenomenon, gastrointestinal (GI) symptoms, lung symptoms, and overall disease severity.
  The HAQ-DI yields a score of 0-3, that indicates the extent of the respondent's functional limitations.
  Each VAS score is scaled from 0 to 3, with 0 being no symptoms and 3 being the worst possible symptom severity.
  A composite VAS score is not created nor are the individual VAS scores incorporated into the HAQ DI score. Typically, each VAS score is reported individually. There is a proposed way to obtain a combined score obtained by pooling the 8 domains of the HAQ DI and the 5 VASs; however, this approach has not yet been widely accepted.
  This is a patient reported outcome.
Change in the diffusing capacity for carbon monoxide (pulmonary function) | 24 and 48 weeks*
  Change in Pulmonary Function as measured by percentage of Improving or worsening DLCO.
  The DLCO (diffusing capacity of the lungs for carbon monoxide) measures the ability of the lungs to transfer gas from inhaled air to the red blood cells in pulmonary capillaries.
  % Improving/worsening DLCO. Analyzed as an ordinal outcome.
  *PFT (pulmonary function test) results will only be analyzed as available under standard of care.
Change in Forced Vital Capacity (pulmonary function) | 24 and 48 weeks*
  Change in Pulmonary Function as measured by percentage of Improving or worsening FVC.
  The FVC (Forced vital Capacity) is the total amount of air exhaled during the FEV (Forced expiratory volume) test.
  % Improving/worsening FVC. Analyzed as an ordinal outcome.
  *PFT (pulmonary function test) results will only be analyzed as available under standard of care.
Combined Response Index in diffuse cutaneous systemic sclerosis score (CRISS) | Baseline (week 0), and at 24, 48 weeks
  To define disease progression
  CRISS score: It is calculated according to changes from the start of a study, compared to an endpoint, by using the modified Rodnan Skin Score (mRSS), the Health Assessment Questionnaire - Disability Index (HAQ-DI), patient and physician global assessment of scleroderma-related health, and forced vital capacity. A CRISS score of ≥ 0.6 indicates likelihood that a patient improved on treatment.
Change in serum concentrations C-Reactive Protein | 12, 24, 36, and 48 weeks
  Change in serum concentrations of the acute phase reactant, CRP
  CRP aids in the evaluation of stress, trauma, infection, inflammation, surgery & associated diseases. Blood levels of C-Reactive Protein (CRP) are known to rise in acute disease to a level of up to 50 mg/L in the presence of slight to moderate inflammatory process. Values >50 mg/L indicate high and extensive inflammatory activity.
Change in serum concentrations of Erythrocyte Sedimentation Rate | 12, 24, 36, and 48 weeks
  Change in serum concentrations of the acute phase reactant, ESR
  Reference ranges:
  Male: 0-10 mm/h Female: 0-20 mm/h
  A faster-than-normal rate may indicate inflammation in the body. Inflammation is part of the immune response system. The higher the number, the higher the likelihood of inflammation.

OTHER OUTCOMES:
Regimen-related toxicities | assessed for duration of treatment up to 48 weeks, and up to 12 weeks post-treatment
  Defined as Adverse Events (AEs) >= Grade 3 and assessed by the investigator as 1 of the following: related or unrelated to treatment.
Infectious complications | assessed for duration of treatment up to 48 weeks, and up to 1 month post-treatment
  Any infectious complication will be tracked under Adverse Event recording
Change in peripheral levels of T-cell activation marker - sIL-2R | 12, 24, 36, and 48 weeks
  interleukin 2 receptor (sIL-2R)
  Serum sIL-2R level is a sensitive and quantitative marker of circulating peripheral blood mononuclear cell activation.
  Normal range of serum sIL-2R is below 2500 pg/ml. High levels may be found in conditions associated with T-cell activation.
Change in peripheral levels of fibrillogenesis - amino terminal propeptide of type III collagen | 12, 24, 36, and 48 weeks
  Changes in serum amino-terminal propeptide of type III collagen levels.
  Amino-terminal propeptide of procollagen type III (PIIINP) is generated during the synthesis of type III collagen. PIIINP is a non-specific marker of soft tissue injury.
  PIIINP in serum has been shown to correlate with fibrillogenesis, and thus to be a potential direct marker of type III collagen deposition.
  PIIINP reference range Adult (>19 years): 1.2 - 4.2 ug/L
  and myofibroblast score in skin biopsies (24 and 48 weeks) if the study looks favorable with respect to potential benefit and safety.
Change in CD30-positive cell count (T-cell marker) in skin biopsies of involved forearm skin | Taken at Baseline (week 0), and 24, 48 weeks
  Measured by immunohistochemistry (IHC) as the percentage of CD30-positive cells per total number of cells/mm2.
  Reference rage not established (there is no range, we are looking for a stat significant change (decrease) from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Janet E Pope, PhD, Principal Investigator — University of Western Ontario, Division of Rheumatology, St. Joseph's Health Care, London, Ontario, Canada
Locations (1):
- Rheumatology Clinic, St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Komocsi A, Vorobcsuk A, Faludi R, Pinter T, Lenkey Z, Kolto G, Czirjak L. The impact of cardiopulmonary manifestations on the mortality of SSc: a systematic review and meta-analysis of observational studies. Rheumatology (Oxford). 2012 Jun;51(6):1027-36. doi: 10.1093/rheumatology/ker357. Epub 2012 Jan 5. PMID 22223705
- [Background] Young A, Khanna D. Systemic sclerosis: a systematic review on therapeutic management from 2011 to 2014. Curr Opin Rheumatol. 2015 May;27(3):241-8. doi: 10.1097/BOR.0000000000000172. PMID 25775190
- [Background] Shah AA, Casciola-Rosen L, Rosen A. Review: cancer-induced autoimmunity in the rheumatic diseases. Arthritis Rheumatol. 2015 Feb;67(2):317-26. doi: 10.1002/art.38928. No abstract available. PMID 25371098
- [Background] Andras C, Ponyi A, Constantin T, Csiki Z, Szekanecz E, Szodoray P, Danko K. Dermatomyositis and polymyositis associated with malignancy: a 21-year retrospective study. J Rheumatol. 2008 Mar;35(3):438-44. Epub 2008 Jan 15. PMID 18203322
- [Background] Hasegawa M, Sato S, Sakai H, Ohashi T, Takehara K. Systemic sclerosis revealing T-cell lymphoma. Dermatology. 1999;198(1):75-8. doi: 10.1159/000018070. PMID 10026408
- [Background] Juarez M, Marshall R, Denton C, Evely R. Paraneoplastic scleroderma secondary to hairy cell leukaemia successfully treated with cladribine. Rheumatology (Oxford). 2008 Nov;47(11):1734-5. doi: 10.1093/rheumatology/ken367. Epub 2008 Sep 23. No abstract available. PMID 18812428
- [Background] Khanna D, Berrocal VJ, Giannini EH, Seibold JR, Merkel PA, Mayes MD, Baron M, Clements PJ, Steen V, Assassi S, Schiopu E, Phillips K, Simms RW, Allanore Y, Denton CP, Distler O, Johnson SR, Matucci-Cerinic M, Pope JE, Proudman SM, Siegel J, Wong WK, Wells AU, Furst DE. The American College of Rheumatology Provisional Composite Response Index for Clinical Trials in Early Diffuse Cutaneous Systemic Sclerosis. Arthritis Rheumatol. 2016 Feb;68(2):299-311. doi: 10.1002/art.39501. PMID 26808827
- [Background] Valentini G, Silman AJ, Veale D. Assessment of disease activity. Clin Exp Rheumatol. 2003;21(3 Suppl 29):S39-41. PMID 12889221
- [Background] Medsger TA Jr, Bombardieri S, Czirjak L, Scorza R, Della Rossa A, Bencivelli W. Assessment of disease severity and prognosis. Clin Exp Rheumatol. 2003;21(3 Suppl 29):S42-6. PMID 12889222
- [Background] Oflazoglu E, Simpson EL, Takiguchi R, Grewal IS, Hanifin JM, Gerber HP. CD30 expression on CD1a+ and CD8+ cells in atopic dermatitis and correlation with disease severity. Eur J Dermatol. 2008 Jan-Feb;18(1):41-9. doi: 10.1684/ejd.2008.0309. Epub 2007 Dec 18. PMID 18086588
- [Background] Clements P, Lachenbruch P, Siebold J, White B, Weiner S, Martin R, Weinstein A, Weisman M, Mayes M, Collier D, et al. Inter and intraobserver variability of total skin thickness score (modified Rodnan TSS) in systemic sclerosis. J Rheumatol. 1995 Jul;22(7):1281-5. PMID 7562759
- [Background] Clements PJ, Lachenbruch PA, Seibold JR, Zee B, Steen VD, Brennan P, Silman AJ, Allegar N, Varga J, Massa M, et al. Skin thickness score in systemic sclerosis: an assessment of interobserver variability in 3 independent studies. J Rheumatol. 1993 Nov;20(11):1892-6. PMID 8308774
- [Background] Furst DE, Khanna D, Mattucci-Cerinic M, Silman AJ, Merkel PA, Foeldvari I; OMERACT 7 Special Interest Group. Scleroderma--developing measures of response. J Rheumatol. 2005 Dec;32(12):2477-80. PMID 16331791
- [Background] Pope JE, Bellamy N. Outcome measurement in scleroderma clinical trials. Semin Arthritis Rheum. 1993 Aug;23(1):22-33. doi: 10.1016/s0049-0172(05)80024-1. PMID 8235663
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180
- [Background] LeRoy EC, Black C, Fleischmajer R, Jablonska S, Krieg T, Medsger TA Jr, Rowell N, Wollheim F. Scleroderma (systemic sclerosis): classification, subsets and pathogenesis. J Rheumatol. 1988 Feb;15(2):202-5. No abstract available. PMID 3361530
- [Background] Sutherland MS, Sanderson RJ, Gordon KA, Andreyka J, Cerveny CG, Yu C, Lewis TS, Meyer DL, Zabinski RF, Doronina SO, Senter PD, Law CL, Wahl AF. Lysosomal trafficking and cysteine protease metabolism confer target-specific cytotoxicity by peptide-linked anti-CD30-auristatin conjugates. J Biol Chem. 2006 Apr 14;281(15):10540-7. doi: 10.1074/jbc.M510026200. Epub 2006 Feb 16. PMID 16484228
- [Background] Ong VH, Denton CP. Innovative therapies for systemic sclerosis. Curr Opin Rheumatol. 2010 May;22(3):264-72. doi: 10.1097/BOR.0b013e328337c3d6. PMID 20190640
- [Background] Becker MO, Bruckner C, Scherer HU, Wassermann N, Humrich JY, Hanitsch LG, Schneider U, Kawald A, Hanke K, Burmester GR, Riemekasten G. The monoclonal anti-CD25 antibody basiliximab for the treatment of progressive systemic sclerosis: an open-label study. Ann Rheum Dis. 2011 Jul;70(7):1340-1. doi: 10.1136/ard.2010.137935. Epub 2010 Nov 10. No abstract available. PMID 21068100
- [Background] Oon S, Huq M, Godfrey T, Nikpour M. Systematic review, and meta-analysis of steroid-sparing effect, of biologic agents in randomized, placebo-controlled phase 3 trials for systemic lupus erythematosus. Semin Arthritis Rheum. 2018 Oct;48(2):221-239. doi: 10.1016/j.semarthrit.2018.01.001. Epub 2018 Jan 6. PMID 29426575
- [Background] Pope J, McBain D, Petrlich L, Watson S, Vanderhoek L, de Leon F, Seney S, Summers K. Imatinib in active diffuse cutaneous systemic sclerosis: Results of a six-month, randomized, double-blind, placebo-controlled, proof-of-concept pilot study at a single center. Arthritis Rheum. 2011 Nov;63(11):3547-51. doi: 10.1002/art.30549. PMID 21769850
- [Background] Gordon JK, Martyanov V, Franks JM, Bernstein EJ, Szymonifka J, Magro C, Wildman HF, Wood TA, Whitfield ML, Spiera RF. Belimumab for the Treatment of Early Diffuse Systemic Sclerosis: Results of a Randomized, Double-Blind, Placebo-Controlled, Pilot Trial. Arthritis Rheumatol. 2018 Feb;70(2):308-316. doi: 10.1002/art.40358. Epub 2017 Dec 29. PMID 29073351
- [Background] Nihtyanova SI, Schreiber BE, Ong VH, Rosenberg D, Moinzadeh P, Coghlan JG, Wells AU, Denton CP. Prediction of pulmonary complications and long-term survival in systemic sclerosis. Arthritis Rheumatol. 2014 Jun;66(6):1625-35. doi: 10.1002/art.38390. PMID 24591477
- [Background] van Laar JM, Farge D, Sont JK, Naraghi K, Marjanovic Z, Larghero J, Schuerwegh AJ, Marijt EW, Vonk MC, Schattenberg AV, Matucci-Cerinic M, Voskuyl AE, van de Loosdrecht AA, Daikeler T, Kotter I, Schmalzing M, Martin T, Lioure B, Weiner SM, Kreuter A, Deligny C, Durand JM, Emery P, Machold KP, Sarrot-Reynauld F, Warnatz K, Adoue DF, Constans J, Tony HP, Del Papa N, Fassas A, Himsel A, Launay D, Lo Monaco A, Philippe P, Quere I, Rich E, Westhovens R, Griffiths B, Saccardi R, van den Hoogen FH, Fibbe WE, Socie G, Gratwohl A, Tyndall A; EBMT/EULAR Scleroderma Study Group. Autologous hematopoietic stem cell transplantation vs intravenous pulse cyclophosphamide in diffuse cutaneous systemic sclerosis: a randomized clinical trial. JAMA. 2014 Jun 25;311(24):2490-8. doi: 10.1001/jama.2014.6368. PMID 25058083
- [Background] Sullivan KM, Goldmuntz EA, Keyes-Elstein L, McSweeney PA, Pinckney A, Welch B, Mayes MD, Nash RA, Crofford LJ, Eggleston B, Castina S, Griffith LM, Goldstein JS, Wallace D, Craciunescu O, Khanna D, Folz RJ, Goldin J, St Clair EW, Seibold JR, Phillips K, Mineishi S, Simms RW, Ballen K, Wener MH, Georges GE, Heimfeld S, Hosing C, Forman S, Kafaja S, Silver RM, Griffing L, Storek J, LeClercq S, Brasington R, Csuka ME, Bredeson C, Keever-Taylor C, Domsic RT, Kahaleh MB, Medsger T, Furst DE; SCOT Study Investigators. Myeloablative Autologous Stem-Cell Transplantation for Severe Scleroderma. N Engl J Med. 2018 Jan 4;378(1):35-47. doi: 10.1056/nejmoa1703327. PMID 29298160
- [Background] Khanna D, Denton CP, Lin CJF, van Laar JM, Frech TM, Anderson ME, Baron M, Chung L, Fierlbeck G, Lakshminarayanan S, Allanore Y, Pope JE, Riemekasten G, Steen V, Muller-Ladner U, Spotswood H, Burke L, Siegel J, Jahreis A, Furst DE. Safety and efficacy of subcutaneous tocilizumab in systemic sclerosis: results from the open-label period of a phase II randomised controlled trial (faSScinate). Ann Rheum Dis. 2018 Feb;77(2):212-220. doi: 10.1136/annrheumdis-2017-211682. Epub 2017 Oct 24. PMID 29066464
- [Background] Namas R, Tashkin DP, Furst DE, Wilhalme H, Tseng CH, Roth MD, Kafaja S, Volkmann E, Clements PJ, Khanna D; Participants in the Scleroderma Lung Study I and members of the Scleroderma Lung Study II Research Group. Efficacy of Mycophenolate Mofetil and Oral Cyclophosphamide on Skin Thickness: Post Hoc Analyses From Two Randomized Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2018 Mar;70(3):439-444. doi: 10.1002/acr.23282. Epub 2018 Feb 9. PMID 28544580
- [Background] Gazi H, Pope JE, Clements P, Medsger TA, Martin RW, Merkel PA, Kahaleh B, Wollheim FA, Baron M, Csuka ME, Emery P, Belch JF, Hayat S, Lally EV, Korn JH, Czirjak L, Herrick A, Voskuyl AE, Bruehlmann P, Inanc M, Furst DE, Black C, Ellman MH, Moreland LW, Rothfield NF, Hsu V, Mayes M, McKown KM, Krieg T, Siebold JR. Outcome measurements in scleroderma: results from a delphi exercise. J Rheumatol. 2007 Mar;34(3):501-9. Epub 2007 Feb 1. PMID 17299843
- [Background] Daoussis D, Melissaropoulos K, Sakellaropoulos G, Antonopoulos I, Markatseli TE, Simopoulou T, Georgiou P, Andonopoulos AP, Drosos AA, Sakkas L, Liossis SN. A multicenter, open-label, comparative study of B-cell depletion therapy with Rituximab for systemic sclerosis-associated interstitial lung disease. Semin Arthritis Rheum. 2017 Apr;46(5):625-631. doi: 10.1016/j.semarthrit.2016.10.003. Epub 2016 Oct 13. PMID 27839742
- [Background] Ramiro S, Sepriano A, Chatzidionysiou K, Nam JL, Smolen JS, van der Heijde D, Dougados M, van Vollenhoven R, Bijlsma JW, Burmester GR, Scholte-Voshaar M, Falzon L, Landewe RBM. Safety of synthetic and biological DMARDs: a systematic literature review informing the 2016 update of the EULAR recommendations for management of rheumatoid arthritis. Ann Rheum Dis. 2017 Jun;76(6):1101-1136. doi: 10.1136/annrheumdis-2016-210708. Epub 2017 Mar 15. PMID 28298374